CLINICAL TRIAL: NCT00361335
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Golimumab, a Fully Human Anti-TNFa Monoclonal Antibody, Administered Intravenously, in Subjects With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: A Study of Safety and Effectiveness of Golimumab in Participants With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR012781; C0524T12 (Other: Centocor, Inc.); 2005-003232-21 (EudraCT Number)
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Golimumab; Methotrexate; Tumor Necrosis Factor-alpha; Immunology
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group I: 2mg/kg Golimumab + MTX (Experimental): Intravenous (IV) infusions of 2mg/kg golimumab at Week 0 and every 12 weeks thereafter with early escape (an additional 2mg/kg IV infusion of golimumab) and dose regimen adjustment (switch to 4mg/kg IV golimumab), depending on joint assessment results, at Week 16 and 24, respectively. The duration of the combined IV treatment period (initial treatment plus early escape and/or dose regimen adjustment) will be a minimum of 48 weeks. The IV treatment period will be followed by the option of subcutaneous (SC) injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, patients will receive methotrexate (MTX) at the same dose as that before study entry
  Interventions: Drug: Golimumab; Drug: Methotrexate
- Group II: 2mg/kg Golimumab only (Experimental): IV infusions of 2mg/kg golimumab at Week 0 and every 12 weeks thereafter with early escape (addition of MTX) and dose regimen adjustment (addition of MTX or switch to 4mg/kg IV golimumab), depending on joint assessment results, at Week 16 and 24, respectively. The duration of the combined IV treatment period (initial treatment plus early escape and/or dose regimen adjustment) will be a minimum of 48 weeks. The IV treatment period will be followed by the option of SC injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, patients will receive placebo (sham MTX) capsules
  Interventions: Drug: Golimumab; Drug: Placebo
- Group III: 4mg/kg Golimumab + MTX (Experimental): IV infusions of 4mg/kg golimumab at Week 0 and every 12 weeks thereafter for a minimum of 48 weeks followed by the option of SC injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, patients will receive MTX at the same dose as that before study entry.
  Interventions: Drug: Golimumab; Drug: Methotrexate
- Group IV: 4mg/kg Golimumab only (Experimental): IV infusions of 4mg/kg golimumab at Week 0 and every 12 weeks thereafter with early escape (addition of MTX) and dose regimen adjustment (addition of MTX), depending on joint assessment results, at Week 16 and 24, respectively. The duration of the combined IV treatment period (initial treatment plus early escape and/or dose regimen adjustment) will be a minimum of 48 weeks. The IV treatment period will be followed by the option of SC injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, patients will receive placebo (sham MTX) capsules.
  Interventions: Drug: Golimumab; Drug: Placebo
- Group V: IV Placebo + MTX (Placebo Comparator): IV infusions of placebo at Week 0 and Week 12 with early escape (switch to 4mg/kg IV golimumab) and dose regimen adjustment (switch to 4mg/kg IV golimumab), depending on joint assessment results, at Week 16 and 24, respectively. The duration of the combined IV treatment period (placebo plus golimumab) will be a minimum of 48 weeks. The IV treatment period will be followed by the option of SC injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition patients will receive MTX at the same dose as that before study entry. Participants still receiving placebo injections at Week 48 are not eligible to enter the Extension Study.
  Interventions: Drug: Methotrexate; Drug: Placebo

INTERVENTIONS:
Drug: Golimumab — 2mg/kg or 4mg/kg will be administered as an IV infusion over 30 minutes
  Arms: Group I: 2mg/kg Golimumab + MTX; Group II: 2mg/kg Golimumab only; Group III: 4mg/kg Golimumab + MTX; Group IV: 4mg/kg Golimumab only
Drug: Methotrexate — Active MTX capsules, filled with microcrystalline cellulose (Avicel PH 102) and a 2.5 mg MTX tablet, will be administered at the same dose as before the study entry.
  Arms: Group I: 2mg/kg Golimumab + MTX; Group III: 4mg/kg Golimumab + MTX; Group V: IV Placebo + MTX
Drug: Placebo — Placebo solution will be administered through IV infusion in Group V and oral placebo capsules (sham MTX) filled with microcrystalline cellulose (Avicel PH 102) will be administered in Group II and IV.
  Other Names: sham MTX
  Arms: Group II: 2mg/kg Golimumab only; Group IV: 4mg/kg Golimumab only; Group V: IV Placebo + MTX

SUMMARY:
The purpose of this study is to assess the clinical effectiveness and safety of golimumab intravenous (IV) infusions every 12 weeks with or without Methotrexate (MTX), compared with MTX alone, in patients with active rheumatoid arthritis (RA) despite concurrent MTX treatment. In addition, the safety of subcutaneous (SC) golimumab injections following transition from IV golimumab infusions will also be evaluated.

DETAILED DESCRIPTION:
This is a Phase III, double blind (neither investigator nor participant knows the treatment received), placebo-controlled (an inactive substance that is compared with the study medication to test whether the study medication has a real effect in clinical study), multicenter, 5-arm (treatment groups) study of golimumab at 2 doses (given with or without MTX over a period of 30 minutes) for at least 48 weeks in patients with active RA despite concurrent MTX therapy. The study consists of a treatment period of golimumab IV infusions (IV Period) which ranges from 48 weeks to approximately 140 weeks, assuming an enrollment period of approximately 92 weeks, and a long-term optional extension period (Extension Study) in which golimumab SC injections will be given for 24 weeks. The end of study will be the time the last participant completes the Week E-40 visit (Extension Study) for safety follow-up assessments. For the IV Period, participants will be randomly assigned to 1 of the 5 treatment groups in a 1:1:1:1:1 ratio (approximately 125 patients per group). At Week 16 and Week 24, joint assessment results will be used to allow participants to enter early escape and dose regimen adjustment, respectively, in a blinded fashion. Treatment will be unblinded after the 48-week database lock and participants will be given the option to participate in the Extension Study and receive SC injections of 50mg golimumab (with or without MTX) every 4 weeks for an additional 24 weeks. Safety will be monitored throughout the study. The entire study duration (IV Period plus Extension Study) for each participant will range from 88 weeks up to 192 weeks, assuming an enrollment period of approximately 92 weeks.

ELIGIBILITY:
Inclusion Criteria:

- Must have a diagnosis of active rheumatoid arthritis (RA) (according to the revised 1987 criteria of the ARA (American Rheumatism Association) with at least 4 swollen and 4 tender joints for at least 3 months prior to screening - Have been treated with and tolerated methotrexate (MTX) at a dose of at least 15 mg per week for at least 3 months prior to screening - Have been on a stable MTX dose of greater than or equal to 15 mg per week and less than or eual to 25 mg per week for at least 4 weeks prior to screening - If using non steroidal anti-inflammatory agents (such as naproxen) or other pain relievers for RA, must be on a stable dose for at least 2 weeks prior to the first administration of study agent

Exclusion Criteria:

- Participants having known hypersensitivity (severe allergy) to human immunoglobulin proteins or other components of golimumab - Having known clinically serious adverse reaction to a biologic anti-TNF agent - Have had history of latent or active granulomatous infection, including tuberculosis, histoplasmosis, or coccidioidomycosis, prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (72):
- United States (20):
  - Peoria, Arizona
  - Aventura, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Voorhees Township, New Jersey
  - Albany, New York
  - Roslyn, New York
  - Charlotte, North Carolina
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Norristown, Pennsylvania
  - West Reading, Pennsylvania
  - Willow Grove, Pennsylvania
  - Amarillo, Texas
  - Fort Worth, Texas
  - Lubbock, Texas
  - Spokane, Washington
- Argentina (6):
  - Buenos Aires
  - Córdoba
  - Rosario
  - San Juan
  - San Miguel de Tucumán
  - Santa Fe
- Australia (6):
  - Fitzroy
  - Heidelberg
  - Maroochydore
  - Melbourne
  - Perth
  - Woodville
- Colombia (4):
  - Barranquilla
  - Bogotá
  - Bucaramanga
  - Floridablanca
- Germany (4):
  - Erlangen
  - Hamburg
  - Magdeburg
  - München
- Hungary (2):
  - Budapest
  - Szolnok
- Latvia (2):
  - Daugavpils
  - Riga
- Lithuania (4):
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
- Malaysia (4):
  - Ipoh
  - Kuching
  - Precinct 7
  - Selangor Darul Ehasan
- Msd06 Gwardiamangia, Malta
- Mexico (4):
  - Colonia del Valle
  - Guadalajara
  - Guadalajara Jalisco
  - Monterrey
- New Zealand (5):
  - Christchurch
  - Dunedin
  - Rotorua
  - Takapuna Auckland
  - Timaru
- Lima, Peru
- Poland (5):
  - Bialystok
  - Elblag
  - Krakow
  - Warsaw
  - Włoszczowa
- Ukraine (4):
  - Kiev
  - Kyiv
  - Symferpol
  - Zhaporizhzhya

REFERENCES:
- [Derived] George MD, Ostergaard M, Conaghan PG, Emery P, Baker DG, Baker JF. Obesity and rates of clinical remission and low MRI inflammation in rheumatoid arthritis. Ann Rheum Dis. 2017 Oct;76(10):1743-1746. doi: 10.1136/annrheumdis-2017-211569. Epub 2017 Jun 12. PMID 28606966
- [Derived] Baker JF, Conaghan PG, Smolen JS, Aletaha D, Shults J, Emery P, Baker DG, Ostergaard M. Development and validation of modified disease activity scores in rheumatoid arthritis: superior correlation with magnetic resonance imaging-detected synovitis and radiographic progression. Arthritis Rheumatol. 2014 Apr;66(4):794-802. doi: 10.1002/art.38304. PMID 24757132
- [Derived] Baker JF, Baker DG, Toedter G, Shults J, Von Feldt JM, Leonard MB. Associations between vitamin D, disease activity, and clinical response to therapy in rheumatoid arthritis. Clin Exp Rheumatol. 2012 Sep-Oct;30(5):658-64. Epub 2012 Oct 17. PMID 22776409
- [Derived] Taylor PC, Ritchlin C, Mendelsohn A, Baker D, Kim L, Xu Z, Mack M, Kremer J. Maintenance of efficacy and safety with subcutaneous golimumab among patients with active rheumatoid arthritis who previously received intravenous golimumab. J Rheumatol. 2011 Dec;38(12):2572-80. doi: 10.3899/jrheum.110570. Epub 2011 Nov 15. PMID 22089463
- [Derived] Kremer J, Ritchlin C, Mendelsohn A, Baker D, Kim L, Xu Z, Han J, Taylor P. Golimumab, a new human anti-tumor necrosis factor alpha antibody, administered intravenously in patients with active rheumatoid arthritis: Forty-eight-week efficacy and safety results of a phase III randomized, double-blind, placebo-controlled study. Arthritis Rheum. 2010 Apr;62(4):917-28. doi: 10.1002/art.27348. PMID 20131276

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 86 investigational sites. The study population included 643 randomized participants from 15 countries.
Pre-assignment Details: A total of 643 participants were randomized in the IV Period (Main Study). A total of 508 participants were randomized in the SC Period (Extension Study); participation in the SC Period was optional.
Groups:
- 2mg/kg Golimumab+ MTX: Participants received intravenous (IV) infusions of 2mg/kg golimumab at Week 0 and every 12 weeks thereafter for a minimum of 48 weeks followed by the option of subcutaneous (SC) injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, participants received methotrexate (MTX) at the same dose as before study entry.
- 2mg/kg Golimumab Only: Participants received IV infusions of 2mg/kg golimumab at Week 0 and every 12 weeks thereafter for a minimum of 48 weeks followed by the option of SC injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, participants received placebo (sham MTX) capsules during the IV Period only.
- 4mg/kg Golimumab + MTX: Participants received IV infusions of 4mg/kg golimumab at Week 0 and every 12 weeks thereafter for a minimum of 48 weeks followed by the option of SC injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, participants received MTX at the same dose as before study entry.
- 4mg/kg Golimumab Only: Participants received IV infusions of 4mg/kg golimumab at Week 0 and every 12 weeks thereafter for a minimum of 48 weeks followed by the option of SC injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, participants received placebo (sham MTX) capsules during the IV Period only.
- IV Placebo + MTX: Participants received IV infusions of placebo at Week 0 and Week 12. At Week 24, depending on joint assessment results (dose regimen adjustment), participants were switched to IV infusions of 4mg/kg golimumab every 12 weeks for a minimum combined treatment period (placebo plus golimumab) of 48 weeks. This was followed by the option of subcutaneous (SC) injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition participants received MTX at the same dose as before study entry. Participants still receiving placebo infusions at Week 48 were not eligible to enter the Extension Study.
- EE/DRA -> 2mg/kg Golimumab + MTX: At Week 16 and Week 24 participants entered early escape (EE) and dose regimen adjustment (DRA), respectively, depending on joint assessment results and received IV infusions of 2mg/kg golimumab (as per protocol) for a minimum combined treatment period (initial treatment plus EE or DRA) of 48 weeks. This was followed by the option of SC injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, participants received MTX at the same dose as before study entry.
- EE/DRA -> 4mg/kg Golimumab + MTX: At Week 16 and Week 24 participants entered EE and DRA, respectively, depending on joint assessment results and received IV infusions of 4mg/kg golimumab (as per protocol) for a minimum combined treatment period (initial treatment plus EE or DRA) of 48 weeks. This was followed by the option of SC injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, participants received MTX at the same dose as before study entry.
Period: IV Period: Baseline to E0
Arm/Group | 2mg/kg Golimumab+ MTX | 2mg/kg Golimumab Only | 4mg/kg Golimumab + MTX | 4mg/kg Golimumab Only | IV Placebo + MTX | EE/DRA -> 2mg/kg Golimumab + MTX | EE/DRA -> 4mg/kg Golimumab + MTX
Started | 129 | 128 | 128 | 129 | 129 | 0 ("0" in column indicates this reporting group is not relevant to the IV Period.) | 0 ("0" in column indicates this reporting group is not relevant to the IV Period.)
Completed | 109 | 99 | 107 | 102 | 105 | 0 | 0
Not Completed | 20 | 29 | 21 | 27 | 24 | 0 | 0
Not completed — Adverse Event | 9 | 4 | 5 | 9 | 8 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Death | 1 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Discontinued oral study agent | 2 | 1 | 1 | 1 | 2 | 0 | 0
Not completed — Protocol-prohibited medications | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Worsening of RA | 0 | 5 | 1 | 4 | 2 | 0 | 0
Not completed — Other | 2 | 9 | 9 | 3 | 2 | 0 | 0
Not completed — Lack of Efficacy | 5 | 9 | 3 | 7 | 8 | 0 | 0
Period: SC Period: Week E0 to Week E24
Arm/Group | 2mg/kg Golimumab+ MTX | 2mg/kg Golimumab Only | 4mg/kg Golimumab + MTX | 4mg/kg Golimumab Only | IV Placebo + MTX | EE/DRA -> 2mg/kg Golimumab + MTX | EE/DRA -> 4mg/kg Golimumab + MTX
Started | 82 (Reporting groups in the SC Period are determined by treatment assignment at Week 24) | 59 (Reporting groups in the SC Period are determined by treatment assignment at Week 24) | 104 (Reporting groups in the SC Period are determined by treatment assignment at Week 24) | 63 (Reporting groups in the SC Period are determined by treatment assignment at Week 24) | 3 (Reporting groups in the SC Period are determined by treatment assignment at Week 24) | 24 (Reporting groups in the SC Period are determined by treatment assignment at Week 24) | 173 (Reporting groups in the SC Period are determined by treatment assignment at Week 24)
Completed | 80 | 56 | 99 | 59 | 3 | 23 | 164
Not Completed | 2 | 3 | 5 | 4 | 0 | 1 | 9
Not completed — Adverse Event | 0 | 2 | 1 | 2 | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Worsening of RA | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 1 | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- 2mg/kg Golimumab+ MTX: Participants received intravenous (IV) infusions of 2mg/kg golimumab at Week 0 and every 12 weeks for a minimum of 48 weeks followed by the option of subcutaneous (SC) injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, participants received methotrexate (MTX) at the same dose as before study entry.
- 4mg/kg Golimumab + MTX: Participants received IV infusions of 4mg/kg golimumab at Week 0 and every 12 weeks for a minimum of 48 weeks followed by the option of SC injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, participants received MTX at the same dose as before study entry.
- 4mg/kg Golimumab Only: Participants received IV infusions of 4mg/kg golimumab at Week 0 and every 12 weeks for a minimum of 48 weeks followed by the option of SC injections of 50mg golimumab every 4 weeks for a further 24 weeks (Extension Study). In addition, participants received placebo (sham MTX) capsules during the IV Period only.
- Total: Total of all reporting groups
Arm/Group | 2mg/kg Golimumab+ MTX | 2mg/kg Golimumab Only | 4mg/kg Golimumab + MTX | 4mg/kg Golimumab Only | IV Placebo + MTX | Total
Number analyzed (Participants) | 129 | 128 | 128 | 129 | 129 | 643
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (11.10) | 49.9 (11.86) | 49.6 (10.96) | 48.4 (12.66) | 50.2 (11.28) | 49.4 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 107 | 103 | 105 | 103 | 517
  Male | 30 | 21 | 25 | 24 | 26 | 126

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an American College of Rheumatology (ACR) 50 Response at Week 14
Description: An ACR 50 response is defined as a greater than or equal to 50 percentage improvement from baseline in: 1. Swollen joint count (66 joints) and tender joint count (68 joints) 2. greater than or equal to 50 percentage improvement in 3 of the following 5 assessments: a. Patient's assessment of pain (VAS) (0-10 cm) b. Patient's Global Assessment of Disease activity (VAS) (0-10 cm) c. Physician's Global Assessment of Disease Activity (VAS) (0-10 cm) d. Patient's assessment of physical function as measured by the Health Assessment Questionnaire (HAQ) e. C reactive protein (CRP).
Time Frame: Week 0 to Week 14
Population: Intent to treat (ITT). Patients considered non-responder if used any pre-specified prohibited medications or discontinued subcutaneous (SC) study agent due to lack of efficacy. Missing ACR components were imputed by Last Observation Carried Forward (LOCF) unless all ACR components are missing in which case considered non-responders.
Measure: Number; unit: Participants
Groups:
- Group I: 2mg/kg Golimumab+ MTX: Participants received intravenous (IV) infusions of 2mg/kg golimumab at Week 0 and every 12 weeks thereafter for a minimum of 48 weeks. In addition, participants received methotrexate (MTX) at the same dose as before study entry.
- Group II: 2mg/kg Golimumab Only: Participants received IV infusions of 2mg/kg golimumab at Week 0 and every 12 weeks thereafter for a minimum of 48 weeks. In addition, participants received placebo (sham MTX) capsules.
- Group III: 4mg/kg Golimumab + MTX: Participants received IV infusions of 4mg/kg golimumab at Week 0 and every 12 weeks thereafter for a minimum of 48 weeks. In addition, participants received MTX at the same dose as before study entry.
- Group IV: 4mg/kg Golimumab Only: Participants received IV infusions of 4mg/kg golimumab at Week 0 and every 12 weeks thereafter for a minimum of 48 weeks. In addition, participants received placebo (sham MTX) capsules.
- Group V: IV Placebo + MTX: Participants received IV infusions of placebo at Week 0 and every 12 weeks thereafter through Week 48. In addition participants received MTX at the same dose as that before study entry.
- Group VI: Combined Groups I and III: Combined Groups I and III (2mg/kg or 4mg/kg Golimumab and Methotrexate)
- Group VII: Combined Groups II and IV: Combined Groups II and IV (2mg/kg or 4mg/kg Golimumab Only)
Arm/Group | Group I: 2mg/kg Golimumab+ MTX | Group II: 2mg/kg Golimumab Only | Group III: 4mg/kg Golimumab + MTX | Group IV: 4mg/kg Golimumab Only | Group V: IV Placebo + MTX | Group VI: Combined Groups I and III | Group VII: Combined Groups II and IV
Number analyzed (Participants) | 129 | 128 | 128 | 129 | 129 | 257 | 257
Participants | 28 | 16 | 27 | 25 | 17 | 55 | 41
Statistical Analysis 1: Comparison: Group V: IV Placebo + MTX vs Group VI: Combined Groups I and III; Hypothesis: Null hypothesis: No difference in ACR 50 response at Wk 14 comparing Groups V vs VI at 0.05 level of significance. Sample size: The sample size of 125 patients in each of the 5 randomized groups will provide at least 90 percentage power to detect a difference in the ACR 50 response rates between groups assuming 13 percentage response in Group V and ~29-31 percentage response in the Group VI at α = 0.05; Test type: Superiority or Other; p = 0.051, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Group I: 2mg/kg Golimumab+ MTX vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in ACR 50 response at Wk 14 comparing Groups I vs V at 0.05 level of significance. Sample size: The sample size of 125 patients in each of the 5 randomized groups will provide at least 90 percentage power to detect a difference in the ACR 50 response rates between groups assuming 13 percentage response in Group V and ~29-31% response in the Group I at α = 0.05; Test type: Superiority or Other; p = 0.073, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Group III: 4mg/kg Golimumab + MTX vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in ACR 50 response at Wk 14 comparing Groups III vs V at 0.05 level of significance. Sample size: The sample size of 125 patients in each of the 5 randomized groups will provide at least 90 percentage power to detect a difference in the ACR 50 response rates between groups assuming 13 percentage response in Group V and ~29-31 percentage response in the Group III at α = 0.05; Test type: Superiority or Other; p = 0.093, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Group V: IV Placebo + MTX vs Group VII: Combined Groups II and IV; Hypothesis: Null hypothesis: No difference in ACR 50 response at Wk 14 comparing Groups VII vs V at 0.05 level of significance. Sample size: The sample size of 125 patients in each of the 5 randomized groups will provide at least 90 percentage power to detect a difference in the ACR 50 response rates between groups assuming 13 percentage response in Group V and ~29-31 percentage response in the Group VII at α = 0.05; Test type: Superiority or Other; p = 0.465, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Group II: 2mg/kg Golimumab Only vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in ACR 50 response at Wk 14 comparing Groups II vs V at 0.05 level of significance. Sample size: The sample size of 125 patients in each of the 5 randomized groups will provide at least 90 percentage power to detect a difference in the ACR 50 response rates between groups assuming 13 percentage response in Group V and ~29-31 percentage response in the Group II at α = 0.05; Test type: Superiority or Other; p = 0.872, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Group IV: 4mg/kg Golimumab Only vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in ACR 50 response at Wk 14 comparing Groups V vs I, V vs III, V vs II, and V vs IV at 0.05 level of significance. Sample size: The sample size of 125 patients in each of the 5 randomized groups will provide at least 90 percentage power to detect a difference in the ACR 50 response rates between groups assuming 13 percentage response in Group V and ~29-31 percentage response in the combined group (I and III) at α = 0.05; Test type: Superiority or Other; p = 0.175, 2-sided Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Participants With an American College of Rheumatology (ACR) 50 Response at Week 24
Description: ACR 50 response is an improvement of greater than or equal to 50 percentage from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (patient's assessment of pain, patient's global assessemnt of disease activity, Physician's global assessment of disease activity (based on a scale of 0=no disease to 10=severe disease), HAQ (20 questions on life activities) and CRP blood test to measure inflammation).
Time Frame: Week 0 to Week 24
Measure: Number; unit: Participants
Arm/Group | Group I: 2mg/kg Golimumab+ MTX | Group II: 2mg/kg Golimumab Only | Group III: 4mg/kg Golimumab + MTX | Group IV: 4mg/kg Golimumab Only | Group V: IV Placebo + MTX | Group VI: Combined Groups I and III | Group VII: Combined Groups II and IV
Number analyzed (Participants) | 129 | 128 | 128 | 129 | 129 | 257 | 257
Participants | 24 | 11 | 32 | 15 | 12 | 56 | 26
Statistical Analysis 1: Comparison: Group V: IV Placebo + MTX vs Group VI: Combined Groups I and III; Null hypothesis: No difference in ACR 50 response at Week 24 comparing Groups V vs VI at 0.05 level of significance; Test type: Superiority or Other; p = 0.002, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Group I: 2mg/kg Golimumab+ MTX vs Group V: IV Placebo + MTX; Null hypothesis: No difference in ACR 50 response at Week 24 comparing Groups I vs V at 0.05 level of significance; Test type: Superiority or Other; p = 0.032, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Group III: 4mg/kg Golimumab + MTX vs Group V: IV Placebo + MTX; Null hypothesis: No difference in ACR 50 response at Week 24 comparing Groups III vs V at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Group V: IV Placebo + MTX vs Group VII: Combined Groups II and IV; Null hypothesis: No difference in ACR 50 response at Week 24 comparing Groups V vs VII at 0.05 level of significance; Test type: Superiority or Other; p = 0.795, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Group II: 2mg/kg Golimumab Only vs Group V: IV Placebo + MTX; Null hypothesis: No difference in ACR 50 response at Week 24 comparing Groups II vs V at 0.05 level of significance; Test type: Superiority or Other; p = 0.844, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Group IV: 4mg/kg Golimumab Only vs Group V: IV Placebo + MTX; Null hypothesis: No difference in ACR 50 response at Week 24 comparing Groups V vs I, V vs III, V vs II, and V vs IV at 0.05 level of significance; Test type: Superiority or Other; p = 0.540, 2-sided Cochran-Mantel-Haenszel

3. Secondary Outcome: Number of Participants With an American College of Rheumatology (ACR) 20 Response at Week 14
Description: ACR 20 response is an improvement of greater than or equal to 20 percentage from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (patient's assessment of pain, patient's global assessemnt of disease activity, Physician's global assessment of disease activity [based on a scale of 0=no disease to 10=severe disease), HAQ (20 questions on life activities] and CRP blood test to measure inflammation).
Time Frame: Week 0 to Week 14
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group I: 2mg/kg Golimumab+ MTX | Group II: 2mg/kg Golimumab Only | Group III: 4mg/kg Golimumab + MTX | Group IV: 4mg/kg Golimumab Only | Group V: IV Placebo + MTX | Group VI: Combined Groups I and III | Group VII: Combined Groups II and IV
Number analyzed (Participants) | 129 | 128 | 128 | 129 | 129 | 257 | 257
Participants | 71 | 51 | 66 | 62 | 36 | 137 | 113
Statistical Analysis 1: Comparison: Group V: IV Placebo + MTX vs Group VI: Combined Groups I and III; Null hypothesis: No difference in ACR 20 response at Wk 14 comparing Groups V vs VI at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Group I: 2mg/kg Golimumab+ MTX vs Group V: IV Placebo + MTX; Null hypothesis: No difference in ACR 20 response at Wk 14 comparing Groups I vs V at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Group III: 4mg/kg Golimumab + MTX vs Group V: IV Placebo + MTX; Null hypothesis: No difference in ACR 20 response at Wk 14 comparing Groups III vs V at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Group V: IV Placebo + MTX vs Group VII: Combined Groups II and IV; Null hypothesis: No difference in ACR 20 response at Wk 14 comparing Groups V vs VII at 0.05 level of significance; Test type: Superiority or Other; p = 0.002, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Group II: 2mg/kg Golimumab Only vs Group V: IV Placebo + MTX; Null hypothesis: No difference in ACR 20 response at Wk 14 comparing Groups II vs V at 0.05 level of significance; Test type: Superiority or Other; p = 0.043, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Group IV: 4mg/kg Golimumab Only vs Group V: IV Placebo + MTX; Null hypothesis: No difference in ACR 20 response at Wk 14 comparing Groups V vs I, V vs III, V vs II, and V vs IV at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, 2-sided Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of Participants With a Disease Activity Index Score 28 (Using C-reactive Protein)Moderate or Good Response at Week 14
Description: DAS28 using CRP is a measure of tender and swollen joints (28 joints each) and the patient's assessment of disease activity. Values range from 0 (best) to 10 (worst). A score of higher than 5.1 indicates high disease activity, and a score below 3.2 indicates low disease activity. A "Good" response is defined as a patient with a DAS28 score of <= 3.2 at Week 14 with improvement from Baseline in DAS28 score of > 1.2. A "Moderate" response is defined as a patient with DAS28 score of >3.2-5.1 at Week 14 with improvement from baseline in DAS28 score of >1.2 or a DAS28 score of <= 5.1 and improvement from baseline in DAS28 score of >0.6 to 1.2
Time Frame: Week 0 to Week 14
Population: Intent to treat. Patients considered non-responder if used any pre-specified prohibited medications or discontinued subcutaneous (SC) study agent due to lack of efficacy. Missing components were imputed by the median component value of all patients in the same stratum unless all components are missing in which case considered non-responders.
Measure: Number; unit: Participants
Arm/Group | Group I: 2mg/kg Golimumab+ MTX | Group II: 2mg/kg Golimumab Only | Group III: 4mg/kg Golimumab + MTX | Group IV: 4mg/kg Golimumab Only | Group V: IV Placebo + MTX | Group VI: Combined Groups I and III | Group VII: Combined Groups II and IV
Number analyzed (Participants) | 129 | 128 | 128 | 129 | 129 | 257 | 257
Participants | 89 | 80 | 94 | 83 | 57 | 183 | 163
Statistical Analysis 1: Comparison: Group V: IV Placebo + MTX vs Group VI: Combined Groups I and III; Hypothesis: Null hypothesis: No difference in DAS28 response using CRP at Wk 14 comparing Groups V vs VI at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Group I: 2mg/kg Golimumab+ MTX vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in DAS28 response using CRP at Wk 14 comparing Groups I vs V at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Group III: 4mg/kg Golimumab + MTX vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in DAS28 response using CRP at Wk 14 comparing Groups III vs V at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Group V: IV Placebo + MTX vs Group VII: Combined Groups II and IV; Hypothesis: Null hypothesis: No difference in DAS28 response using CRP at Wk 14 comparing Groups V vs VII at 0.05 level of significance; Test type: Superiority or Other; p < 0.001, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Group II: 2mg/kg Golimumab Only vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in DAS28 response using CRP at Wk 14 comparing Groups II vs V at 0.05 level of significance; Test type: Superiority or Other; p = 0.003, 2-sided Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Group IV: 4mg/kg Golimumab Only vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in DAS28 response using CRP at Wk 14 comparing Groups V vs I, V vs III, V vs II, and V vs IV at 0.05 level of significance; Test type: Superiority or Other; p = 0.001, 2-sided Cochran-Mantel-Haenszel; No adjustments were made to control for multiplicity

5. Secondary Outcome: Physical Component Summary (PCS) Score of the Short Form-36 (SF-36) at Week 14
Description: The SF-36 consists of 8 multi-item scales: limitations in physical functioning due to health problems, usual role activities due to physical health problems, bodily pain, usual role activities due to personal or emotional problems, social functioning due to physical or mental health problems, general mental health (psychological distress and well-being), vitality and general health perception. The values are 100=best to 0=worst.
Time Frame: Weeks 0 to Week 14
Population: Intent to treat (ITT). Missing components were imputed by the median component value of all patients in the same Stratum at baseline, and last observation carried forward (LOCF) at Week 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group I: 2mg/kg Golimumab+ MTX | Group II: 2mg/kg Golimumab Only | Group III: 4mg/kg Golimumab + MTX | Group IV: 4mg/kg Golimumab Only | Group V: IV Placebo + MTX | Group VI: Combined Groups I and III | Group VII: Combined Groups II and IV
Number analyzed (Participants) | 129 | 128 | 128 | 129 | 129 | 257 | 257
Units on a scale | 6.92 (9.175) | 4.03 (7.462) | 6.76 (8.252) | 5.14 (9.674) | 4.27 (7.216) | 6.84 (8.702) | 4.58 (8.644)
Statistical Analysis 1: Comparison: Group V: IV Placebo + MTX vs Group VI: Combined Groups I and III; Hypothesis: Null hypothesis: No difference in change from baseline in PCS score of SF-36 at Wk 14 comparing Groups V vs VI at 0.05 level of significance; Test type: Superiority or Other; p = 0.005, 2-sided ANOVA on van der Waerden
Statistical Analysis 2: Comparison: Group I: 2mg/kg Golimumab+ MTX vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in change from baseline in PCS score of SF-36 at Wk 14 comparing Groups I vs V at 0.05 level of significance; Test type: Superiority or Other; p = 0.014, 2-sided ANOVA on van der Waerden
Statistical Analysis 3: Comparison: Group III: 4mg/kg Golimumab + MTX vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in change from baseline in PCS score of SF-36 at Wk 14 comparing Groups III vs V at 0.05 level of significance; Test type: Superiority or Other; p = 0.014, 2-sided ANOVA on van der Waerden
Statistical Analysis 4: Comparison: Group I: 2mg/kg Golimumab+ MTX vs Group VII: Combined Groups II and IV; Hypothesis: Null hypothesis: No difference in change from baseline in PCS score of SF-36 at Wk 14 comparing Groups I and VII at 0.05 level of significance; Test type: Superiority or Other; p = 0.996, 2-sided ANOVA on van der Waerden
Statistical Analysis 5: Comparison: Group II: 2mg/kg Golimumab Only vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in change from baseline in PCS score of SF-36 at Wk 14 comparing Groups II vs V at 0.05 level of significance; Test type: Superiority or Other; p = 0.738, 2-sided ANOVA on van der Waerden
Statistical Analysis 6: Comparison: Group IV: 4mg/kg Golimumab Only vs Group V: IV Placebo + MTX; Hypothesis: Null hypothesis: No difference in change from baseline in PCS score of SF-36 at Wk 14 comparing Groups V vs I, V vs III, V vs II, and V vs IV at 0.05 level of significance; Test type: Superiority or Other; p = 0.788, 2-sided ANOVA on van der Waerden — No adjustments were made to control for multiplicity

ADVERSE EVENTS:
Time Frame: IV Period: Baseline through Week 48 for all participants, and up to the start of the SC Period (Week E0) for participants who opted to enter the SC Period (Extension Study). SC Period: Week E0 through Week E40.
Description: The number of participants reported at risk for AEs in each treatment (tx) group is based on actual tx received during the study and may differ from the number of participants who started tx in the study. Participants may be counted more than once in the analysis of AEs if they received tx at more than one dose level in the study.
Groups:
- IV Period: 2mg/kg Golimumab+ MTX: Participants who received 2mg/kg IV golimumab and methotrexate (MTX). Follow-up time was counted in this treatment group until the participant started to receive 4mg/kg IV golimumab. Participants may have missed one or more golimumab and/or MTX doses. Participants must have received MTX at some point while receiving 2mg/kg IV golimumab and before receiving 4mg/kg IV golimumab
- IV Period: 2mg/kg Golimumab Only: Participants who received 2mg/kg IV golimumab only. Follow-up time was counted in this treatment group until the participant started to receive 4mg/kg IV golimumab. Participants may have missed one or more golimumab doses. Participants must not have received any MTX while receiving 2mg/kg IV golimumab.
- IV Period: 4mg/kg Golimumab + MTX: Participants who received at least one 4 mg/kg IV golimumab dose and MTX. Follow-up time was counted in this treatment group from the first 4mg/kg IV golimumab infusion. Participants may have missed one or more golimumab and/or MTX doses. Participants must have received MTX at some point while receiving 4mg/kg IV golimumab.
- IV Period: 4mg/kg Golimumab Only: Participants who received at least one 4mg/kg IV golimumab dose. Follow-up time was counted in this treatment group from the first 4mg/kg IV golimumab infusion. Participants may have missed one or more golimumab doses. Participants must not have received any MTX while receiving 4mg/kg IV golimumab.
- IV Period: Placebo + MTX: Participants who received IV placebo and MTX only. Follow-up time was counted in this group until the participant started to receive IV golimumab.
- SC Period: 50mg Golimumab + MTX: Participants who received 50mg SC golimumab and MTX.
- SC Period: 50mg Golimumab Only: Participants who received 50mg golimumab only. Participants must not have received any MTX while receiving 50mg SC golimumab.
Arm/Group | IV Period: 2mg/kg Golimumab+ MTX | IV Period: 2mg/kg Golimumab Only | IV Period: 4mg/kg Golimumab + MTX | IV Period: 4mg/kg Golimumab Only | IV Period: Placebo + MTX | SC Period: 50mg Golimumab + MTX | SC Period: 50mg Golimumab Only
Serious Adverse Events (participants affected / at risk) | 25/182 | 17/128 | 47/336 | 8/127 | 7/129 | 38/419 | 8/117
Other Adverse Events (participants affected / at risk) | 109/182 | 71/128 | 190/336 | 70/127 | 65/129 | 94/419 | 26/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Period: 2mg/kg Golimumab+ MTX (N=182) | IV Period: 2mg/kg Golimumab Only (N=128) | IV Period: 4mg/kg Golimumab + MTX (N=336) | IV Period: 4mg/kg Golimumab Only (N=127) | IV Period: Placebo + MTX (N=129) | SC Period: 50mg Golimumab + MTX (N=419) | SC Period: 50mg Golimumab Only (N=117)
Pneumonia (Infections and infestations) | 1 | 3 | 3 | 1 | 1 | 5 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 4 | 0 | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye abcess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Complicated fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ovarian low malignant potential tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Syringomyelia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Generalized anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine cervical squamous metaplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anogenital warts (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymph node tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendix disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intevertebral discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Narcotic intoxication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervical cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Period: 2mg/kg Golimumab+ MTX (N=182) | IV Period: 2mg/kg Golimumab Only (N=128) | IV Period: 4mg/kg Golimumab + MTX (N=336) | IV Period: 4mg/kg Golimumab Only (N=127) | IV Period: Placebo + MTX (N=129) | SC Period: 50mg Golimumab + MTX (N=419) | SC Period: 50mg Golimumab Only (N=117)
Upper respiratory tract infection (Infections and infestations) | 22 | 14 | 41 | 16 | 12 | 30 | 10
Bronchitis (Infections and infestations) | 14 | 10 | 26 | 8 | 7 | 22 | 2
Nasopharyngitis (Infections and infestations) | 13 | 9 | 13 | 8 | 7 | 19 | 9
Influenza (Infections and infestations) | 6 | 10 | 10 | 5 | 1 | 15 | 3
Urinary tract infection (Infections and infestations) | 8 | 5 | 21 | 7 | 2 | 7 | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 12 | 20 | 19 | 12 | 6 | 29 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 6 | 20 | 6 | 7 | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 15 | 4 | 14 | 7 | 2 | 15 | 4
Nausea (Gastrointestinal disorders) | 20 (129) | 4 (128) | 36 (128) | 7 (129) | 9 (129) | 10 | 1
Dyspepsia (Gastrointestinal disorders) | 12 | 3 | 17 | 4 | 2 | 6 | 0
Vomiting (Gastrointestinal disorders) | 8 | 2 | 11 | 4 | 8 | 6 | 2
Headache (Nervous system disorders) | 17 | 8 | 26 | 8 | 13 | 20 | 2
Rash (Skin and subcutaneous tissue disorders) | 8 | 9 | 9 | 6 | 2 | 5 | 2
Hypertension (Vascular disorders) | 14 | 8 | 15 | 4 | 5 | 7 | 1
Alanine aminotransferase increased (Investigations) | 15 | 3 | 19 | 3 | 8 | 18 | 3
Aspartate aminotransferase increased (Investigations) | 7 | 1 | 11 | 0 | 8 | 10 | 3
Sinusitis (Infections and infestations) | 11 | 3 | 24 | 7 | 6 | 15 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 18 | 5 | 5 | 7 | 2

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse events (NAE) excludes patients who only had NAE that occurred in <=5% of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.